CLINICAL TRIAL: NCT03367325
Title: A New Clinical Decision Support Tool for Improving the Adequacy of Anticoagulant Therapy and Reduce Stroke Incidence in Non-valvular Atrial Fibrillation: a Randomized Clinical Trial in Primary Care
Brief Title: Clinical Decision Support Tool for Improving the Adequacy of Anticoagulant Therapy in Non-valvular Atrial Fibrillation
Acronym: NACOs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Institut Català de la Salut (Other); Department of Health, Generalitat de Catalunya (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SLT002/16/00146
Record Dates: First submitted 2017-11-20; First posted 2017-12-08 (Actual); Last update posted 2018-12-21 (Actual); Status verified 2018-12

CONDITIONS: Atrial Fibrillation; Anticoagulants; Clinical Decision Support Systems
Keywords: non-valvular atrial fibrillation; time in therapeutic range; primary care
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CDS-NVAF benefiting group (Experimental): CDS-NVAF = Clinical decision support (CDS) tool for improving the adequacy of the anticoagulant therapy adequacy in non-valvular atrial fibrillation (NVAF)
  Interventions: Device: CDS-NVAF
- CDS-NVAF not-benefiting group (No Intervention)

INTERVENTIONS:
Device: CDS-NVAF — The CDS-NVAF is intended for patients diagnosed with NVAF and treated with VKA. This tool calculates the time in the therapeutic range (TTR) using the Rosendaal method considering the last International Normalized Ratio (INR) data. The INR data are found in the clinical history of NVAF patients. The CDS-NVAF will be activated when the physician introduces the last INR value. At this time the TTR will be calculated automatically. If the TTR value is < 65%, a pop up screen with a warning text will open suggesting a change to DOAC therapy. The physician can decide whether to change or not the previous prescription. If the TTR value in > 65% the pop up screen will not appear. The TTR value will remain registered on the screen of the follow up of oral anticoagulant use and can be consulted in future queries. The diffusion of the CDS-NVAF will be made by an announcement on the first day of the intervention when the health care professional opens the electronic clinical history.
  Arms: CDS-NVAF benefiting group

SUMMARY:
Atrial fibrillation (AF) is the most common cardiac arrhythmia and increases the risk of ischemic stroke 4-5-fold. The prevention of complications is based on oral or antiplatelet anticoagulant treatment. The first choice of anticoagulant therapy (AT) is the vitamin K antagonist (VKA). Contraindication to VKA or poor control of the International Normalized Ratio leads to the administration of direct-acting oral anticoagulants (DOACs). There is a trend towards inadequate AT in non-valvular AF (NVAF) patients.

The Objective of the study is evaluate the impact of the implementation of a decision support tool linked to digital clinical history on the adequacy of AT, the incidence of complications and the mortality in patients with NVAF in primary health care of the Catalan Institute of Health (ICS).

ELIGIBILITY:
Inclusion Criteria (all criteria must be met):

* Patients diagnosed with NVAF one year prior to the implementation of the computerized tool;
* Patients receiving anticoagulant treatment with DOACs or VKAs;
* Patients followed in primary care (with at least 6 INR controls during the year prior to the intervention).

Exclusion Criteria:

* Patients with INR control in the reference hospital;
* patients with valvular AF (mitral stenosis);
* patients with a prosthetic heart valve;
* change to another primary care center.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63001 (Estimated)
Dates: Start 2017-12-15 (Actual); Primary Completion 2019-12-15 (Estimated); Study Completion 2019-12-15 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of Thromboembolic events | Two years after the beginning of the intervention
  Thromboembolic events: acute myocardial infarction or angina, ischemic stroke, peripheral embolism or transient ischemic attack (TIA)
Incidence rate of Hemorrhagic events | Two years after the beginning of the intervention
  Hemorrhagic events: intracranial hemorrhage and gastrointestinal hemorrhage
Incidence rate of mortality | Two years after the beginning of the intervention
  All-cause mortality
Adequacy of anticoagulant treatment | one year after the beginning of the intervention
  This variable encompasses the adequacy of the anticoagulant treatment, taking into account if an adequate change has occurred or not.
  0 = No adequate change (when an inadequate change has been produced or when an inadequate treatment has been maintained)
  1 = adequate change (when an adequate change has been produced or when an adequate treatment has been maintained) The adequacy of the anticoagulant therapy in patients with NVAF will be based on the fulfillment of the criteria of the Ministry of Health, Social Services and Equality of Spain, 2016*
  * Ministry of Health, Social Services and Equality. Criteria and recommendations for the use of direct oral anticoagulants (ACOD) in the prevention of stroke and systemic embolism in patients with non-valvular atrial fibrillation. 2016. available in: https://www.aemps.gob.es/medicamentosUsoHumano/informesPublicos/docs/criterios-anticoagulantes-orales.pdf

SECONDARY OUTCOMES:
Sociodemographic characteristics of the patients | at the beginning of the intervention
  age, sex, primary care area assigned, physician assigned
Primary Care Center (PCC) characteristics: teaching center | at the beginning of the intervention
  This variable encompasses if a PCC is a teaching center or not
Primary Care Center (PCC) characteristics: urban/rural | at the beginning of the intervention
  This variable encompasses if a PCC is located at urban o rural area
Primary Care Center (PCC) characteristics: socioeconomic deprivation index (MEDEA) | at the beginning of the intervention
  This variable encompasses the socioeconomic deprivation index (MEDEA) of each PCC
Primary Care Center (PCC) characteristics: Standard of Health Care Quality (SHCQ) | at the beginning of the intervention
  This variable encompasses the Standard of Health Care Quality of each PCC
Primary Care Center (PCC) characteristics: Standard of Quality of Pharmaceutical Prescription (SQPP) | at the beginning of the intervention
  This variable encompasses the Standard of Quality of Pharmaceutical Prescription of each PCC
Characteristics of the professional: age | at the beginning of the intervention
  This variable encompasses the age of the professional
Characteristics of the professional: sex | at the beginning of the intervention
  This variable encompasses the sex of the professional
Characteristics of the professional: PCC | at the beginning of the intervention
  This variable identifies the PCC of the professional
Characteristics of the professional: type of work contract | at the beginning of the intervention
  This variable encompasses the type of work contract of the professional
Characteristics of the professional: Standard of Health Care Quality (SHCQ) | at the beginning of the intervention
  This variable encompasses the Standard of Health Care Quality of the professional
Characteristics of the professional: Standard of Quality of Pharmaceutical Prescription (SQPP) | at the beginning of the intervention
  This variable encompasses the Standard of Quality of Pharmaceutical Prescription of the professional
Treatment by direct-acting oral antagonists | at the beginning of the intervention and one year after the beginning of the intervention
  Direct-acting oral antagonists: dabigatran, apixaban or rivaroxaban
Treatment by Vitamin K antagonists | at the beginning of the intervention and one year after the beginning of the intervention
  Vitamin K antagonists: acenocoumarol or warfarin
Treatment by heparin | at the beginning of the intervention and one year after the beginning of the intervention
  presence / absence of heparin treatment
Thromboembolic risk CHA2DS2-VASC (congestive heart failure, hypertension, age 75 years or older, diabetes mellitus, previous stroke or transient ischemic attack, vascular disease, age 65 to 74 years, female) score | at the beginning of the intervention and one year after the beginning of the intervention
  The score indicates the risk of a patient with non-valvular atrial fibrillation of suffering a stroke in one year. The score goes from 0 (absence of risk) to 10 (greater risk).
Bleeding risk HAS-BLED (Hypertension, Abnormal liver/renal function, Stroke, Bleeding history or predisposition, Labile INR, Elderly (>65 years), and Drugs/alcohol) score | at the beginning of the intervention and one year after the beginning of the intervention
  The score allows the calculation of the risk of bleeding in patients with non-valvular atrial fibrillation receiving oral anticoagulant treatment based on the risk factors associated with the probability of bleeding.
  0 = low risk; 1 = intermediate risk; 2 = intermediate risk; ≥3 = high risk

CONTACTS AND LOCATIONS:
Locations (1):
- Fundació Institut Universitari per a la recerca a l'Atenció Primària de Salut Jordi Gol i Gurina (IDIAPJGol), Barcelona, Spain

REFERENCES:
- [Derived] Dalmau Llorca MR, Aguilar Martin C, Carrasco-Querol N, Hernandez Rojas Z, Rodriguez Cumplido D, Castro Blanco E, Queiroga Goncalves A, Fernandez-Saez J, Perez-Villacastin J. Clinical value of a tool for managing oral anticoagulation in nonvalvular atrial fibrillation in primary health care. Randomized clinical trial. Rev Esp Cardiol (Engl Ed). 2024 Jun;77(6):471-480. doi: 10.1016/j.rec.2023.11.009. Epub 2023 Dec 4. English, Spanish. PMID 38056770
- [Derived] Dalmau Llorca MR, Goncalves AQ, Forcadell Drago E, Fernandez-Saez J, Hernandez Rojas Z, Pepio Vilaubi JM, Rodriguez Cumplido D, Morral Parente RM, Aguilar Martin C. A new clinical decision support tool for improving the adequacy of anticoagulant therapy and reducing the incidence of stroke in nonvalvular atrial fibrillation: A randomized clinical trial in primary care. Medicine (Baltimore). 2018 Jan;97(3):e9578. doi: 10.1097/MD.0000000000009578. PMID 29504981